CLINICAL TRIAL: NCT03625401
Title: A Pilot, Phase 2a, Multi-Center, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Investigate the Safety and Tolerability, Efficacy, and Pharmacokinetics of AD-35 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety of AD-35 in Treatment of Subjects With Mild to Moderate Alzheimer's Disease
Acronym: ROAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hisun-AD-35-003
Record Dates: First submitted 2018-07-24; First posted 2018-08-10 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: mild to moderate
MeSH Terms: conditions — Alzheimer Disease | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: AD-35 60 mg group: 2 AD-35 30 mg tablets and 1 placebo tablet; Placebo group: 3 placebo tablets.
Who Masked: Participant, Investigator
Masking Description: During the double-blind period, all of the study personnel, including Investigators, site personnel,the Sponsor's staff (eg, clinical research associate [CRA]/monitor), and study subjects will be blinded to treatment assignment. Placebo and AD-35 will be identical in appearance and packaging to preserve blinding.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AD-35 60 mg (Experimental): AD-35 60 mg group: 2 AD-35 30 mg tablets and 1 placebo tablet
  Interventions: Drug: AD-35 60mg group
- Placebo of AD-35 30 mg (Placebo Comparator): Placebo group: 3 placebo tablets
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: AD-35 60mg group — AD-35 60mg QD
  Arms: AD-35 60 mg
Drug: Placebo group — Placebo: 3 placebo of AD-35 30mg tablets
  Arms: Placebo of AD-35 30 mg

SUMMARY:
multi-center, randomized, double-blind, parallel-group,placebo-controlled study to evaluate the safety and tolerability, efficacy, and PK of 60 mg AD-35 administered QD during 6 months of double-blind treatment followed by a second 6 months of open-label treatment to subjects with mild to moderate AD.

DETAILED DESCRIPTION:
Approximately 55 subjects are planned to be enrolled for the entire study. Subjects will be randomized on Day 1 via a centralized interactive response technology (IRT) in a 1:2 ratio to receive placebo or 60 mg AD-35. The Data Safety Monitoring Board (DSMB) will review safety information after the first 30 subjects have completed the Day 30 Visit and make any necessary recommendations regarding changes to the conduct of the study.

After the first 6 months of double-blind treatment, subjects initially on placebo will transition to active study drug, and all subjects will receive 60 mg AD-35 for an additional 6 months of open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be diagnosed with probable AD in accordance with the National Institute on Aging and Alzheimer's Association (NIA-AA) (2011) criteria.
2. Subjects must have a Mini-Mental State Examination (MMSE) score of ≥15 and ≤26 at screening and baseline.
3. Subjects must have a brain magnetic resonance imaging (MRI) scan that is consistent with a clinical diagnosis of probable AD.
4. Subjects should not have received Aβ-based or tau-based treatment for AD.
5. Subjects who were previously treated with Acetyl cholinesterase inhibitor (AChEI) or memantine, must have been off of the therapy for at least 3 months prior to baseline assessments. Subjects who have been taking AChEI or memantine for ≤7 days may be considered for enrollment in this study.
6. For subjects who are currently receiving other non-excluded prescription or over-the-counter medications that might affect cognitive function (eg, non-anticholinergic antidepressants, atypical antipsychotics, non-benzodiazepine anxiolytics, soporifics, centrally acting anticholinergic antihistamines, centrally acting anticholinergic antispasmodics):

   * Treatment must be at a stable dose for ≥1 month prior to randomization and throughout the duration of the study.
   * Treatment given intermittently and on a short-term basis must not be administered within 5 half-lives prior to the screening of neurocognitive assessments.
7. Subjects must be male or female between 50 years to 85 years of age (inclusive), at screening.
8. Female subjects must be post-menopausal for at least 2 consecutive years or surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 6 months prior to screening.
9. Male subjects with partners of reproductive potential must agree to use a reliable means of contraception (eg, minimum condom + spermicide) during the study and 30 days after discontinuing the study drug.
10. Subjects must have a reliable caregiver with contact at least 3 times per week (combination of face to face visits and telephone contact acceptable). The caregiver must be able to oversee the subject's compliance with study drug and participate in the subject's clinical assessment, to provide meaningful input into the NPI, ADCS-ADL, and CIBIC+.
11. Subjects (or subject's legally authorized representatives and their caregivers) must be able to provide informed consent.
12. Subjects (and their caregivers) must be able to read, write, speak, and understand English to ensure compliance with cognitive testing and study visit procedures.
13. Subjects (and their caregivers) must be willing and able to comply with the protocol's requirements.
14. Subjects must weigh between 45 kg and 90 kg (inclusive), at screening.
15. Subjects must be in general good health in the opinion of the Investigator, based on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) in triplicate, and clinical laboratory values.

Exclusion Criteria:

1. Lack of peripheral venous access.
2. Uncorrected impairment of vision or hearing that would preclude the subject from taking tests, or subjects lacking the ability to communicate.
3. Inability to tolerate MRI procedures or contraindication to MRI, including but not limited to MRI incompatible pacemakers; implantable cardioverter defibrillators; cochlear implants; cerebral aneurysm clips; implanted infusion pumps; implanted nerve stimulators; metallic splinters in the eye; other magnetic, electronic, or mechanical implants; or any other clinical history or examination finding that, in the judgment of the Investigator, would pose a potential hazard in combination with MRI.
4. Severe or unstable medical condition that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to complete the study assessments.
5. History or presence of clinically evident vascular disease potentially affecting the brain (eg, stroke, clinically significant carotid or vertebral stenosis or plaque, aortic aneurysm, intracranial aneurysm, cerebral hemorrhage, arteriovenous malformation).
6. History of severe, clinically significant (persistent neurologic deficit or structural brain damage) central nervous system trauma (eg, cerebral contusion).
7. History or presence of intracranial tumor (eg, meningioma, glioma).
8. Presence of infections that affect the brain function or history of infections that resulted in neurologic sequelae (eg, syphilis, neuroborreliosis, viral or bacterial meningitis/encephalitis,human immunodeficiency virus encephalopathy).
9. History or presence of systemic autoimmune disorders potentially causing progressive neurologic disease (eg, multiple sclerosis, lupus erythematosus, anti-phospholipid antibody syndrome, Behçet disease).
10. History or presence of psychiatric disease other than AD that may affect cognition or prevent completion of study procedures, including but not limited to clinically significant major psychiatric disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) (eg, major depression, schizophrenia, bipolar disorder).

    • A history of major depression is acceptable if no episode has been reported within the previous 5 years.
11. History or presence of a neurologic disease other than AD that may affect cognition, including but not limited to Parkinson's disease, corticobasal degeneration, dementia with Lewy bodies, Creutzfeldt-Jakob disease, progressive supranuclear palsy, frontotemporal degeneration, Huntington's disease, normal pressure hydrocephalus, and hypoxia.
12. History of seizures with the exception of childhood febrile seizures.
13. Known or suspected history of alcohol or drug abuse within the previous 5 years (DSM-V criteria).
14. Evidence of malignancies, acute infections, renal failure that requires dialysis, or other unstable medical disease not related to AD that in the Investigator's opinion would preclude subject participation.

    • This does not include any cancer (except adequately treated basal or squamous cell skin cancer) that is not being actively treated with anti-cancer drugs or radiotherapy as well as cancers that are considered to have low probability of recurrence (with supporting documentation of this from the treating oncologist, if possible).
15. History or presence of atrial fibrillation that poses a risk for future stroke in the Investigator's judgment.
16. Severe heart disease (history of myocardial infarction, congestive heart disease, history of unstable angina pectoris, clinically significant ECG abnormality) within 6 months prior to screening. Subjects with peripheral arterial disease will not be excluded if they are stable for at least 6 months prior to screening.
17. Clinically significant vital signs, laboratory, or ECG abnormalities (eg, abnormally prolonged or shortened heart rate, clinical significant arrhythmias, corrected QT interval [QTcF] >450 ms) in the Investigator's judgement. ECG abnormalities should be confirmed by Investigator based on the central read results provided by the ECG core laboratory (Medpace Cardiovascular Core Laboratory [MCCL]).
18. Subjects must not have an estimated glomerular filtration rate of <30 mL/min/1.73 m2, at screening.
19. Impaired hepatic function, as indicated by transaminases >2 times the upper limit of normal or abnormalities in synthetic function tests judged by the Investigator to be clinically significant.
20. Evidence of poorly-controlled diabetes (glycosylated hemoglobin >8.0%).
21. Presence of superficial siderosis of central nervous system, or >4 cerebral microhemorrhages, or evidence of a prior cerebral macrohemorrhage as assessed by T2*-weighted gradient-recalled-echo (GRE) MRI.
22. Presence of significant cerebral vascular pathology as assessed by MRI.
23. Treatment with any investigational agent within 5 half-lives or 4 weeks prior to screening, whichever is longer.
24. Cognitive dysfunction that might be due to past or current medication (eg, chemotherapy, steroids).
25. Treatment with any biologic therapy within 5 half-lives or 3 months prior to screening, whichever is longer, or any subject who has been in an Alzheimer Aβ or tau vaccination trial unless known to have received only placebo.
26. Treatment with anticholinergic antidepressants, typical antipsychotics, or barbiturates.
27. Chronic use of opiates, opioids, or benzodiazepines:

    • Intermittent short-term use is allowed except within 5 half-lives prior to any neurocognitive assessment.
28. Use or intention to use any medications/products that are cytochrome P450 (CYP)3A4 substrates with narrow therapeutic indexes.
29. Use or intention to use any medications/products that are known to be strong inducers/inhibitors of CYP3A4 within 7 days prior to the first dose and throughout the period of study drug administration.
30. Consumption of grapefruit juice or grapefruit-containing products within 7 days prior to the first dose and throughout the period of study drug administration.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
ADAS-cog 11 score | The primary efficacy endpoint will be change in the ADAS-cog 11 score from baseline to 6 months.
  The ADAS-cog 11 score is a 70-point scale administered by a clinician and is a standard measure to assess change in cognitive function in subjects with mild to moderate AD

SECONDARY OUTCOMES:
NPI score | The secondary efficacy endpoint will be the change from baseline in the NPI score at 6 and 12 months
  NPI score identifies any changes for cognition, behavior, and global function and provide a measure of overall clinical improvement
ADCS-ADL score | The secondary efficacy endpoint will be the change from baseline in the ADCS-ADL score at 6 and 12 months
  ADCS-ADL score identifies any changes for cognition, behavior, and global function and provide a measure of overall clinical improvement
CIBIC+ score | The secondary efficacy endpoint will be the change from baseline in the CIBIC+ score at 6 and 12 months
  CIBIC+ score identifies any changes for cognition, behavior, and global function and provide a measure of overall clinical improvement
ADAS-cog 11 score | The secondary efficacy endpoint will be the change from baseline in ADAS-cog 11 score at 12 months
  The ADAS-cog 11 score is a 70-point scale administered by a clinician and is a standard measure to assess change in cognitive function in subjects with mild to moderate AD

CONTACTS AND LOCATIONS:
Overall Officials: Rentian (Roy) Feng, PhD, Study Director — Zhejiang Hisun Pharmaceuticals Co., Ltd
Locations (10):
- United States (10):
  - Northern California Research, Sacramento, California
  - Pacific Research Network, Inc., San Diego, California
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Meridien Research, Maitland, Florida
  - Meridien Research, Spring Hill, Florida
  - NeuroStudies, Decatur, Georgia
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Clinilabs, Inc., New York, New York